CLINICAL TRIAL: NCT05166135
Title: Real-world Study in Acute Leukemia: Epidemiology, Treatment Patterns and Outcomes for B-cell ALL and AML in Adult Patients From Latin America - LOYAL Study
Brief Title: Latin American Real-world Study in Acute Leukemia
Acronym: LOYAL
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001302; LOYAL (Other: Alias Study Number)
Record Dates: First submitted 2021-11-10; First posted 2021-12-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia
Keywords: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Relapsed Refractory B-cell Acute Lymphoblastic Leukemia; Acute Leukemia in Latin America; LOYAL study
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Myeloid Leukemia: Patients ≥18 years old at diagnosis, with de novo AML diagnosed between 01 January 2015 and 31 December 2019, as documented in the medical chart and according to the physician's notes, and with at least 1 line of treatment for AML within the study period.
- Relapsed/Refractory Acute Lymphoid Leukemia: Patients ≥18 years old at diagnosis, with R/R ALL diagnosed between 01 January 2015 and 31 December 2019, as documented in the medical chart and according to the physician's notes, and with at least 1 line of treatment for R/R ALL within the study period.

SUMMARY:
The objective of the study is to describe the current epidemiology, treatment patterns, outcomes and healthcare resource use of adult patients diagnosed with relapsed/refractory (R/R) B-cell ALL and de novo AML in 4 Latin American countries.

DETAILED DESCRIPTION:
This is a retrospective multicenter non-interventional study using real-world data collected from medical records of newly diagnosed AML or with relapsed/refractory B-cell ALL diagnosed between 01 January 2015 and 31 December 2019 in 4 Latin American countries: Argentina, Brazil, Chile, and Colombia. In addition, as secondary objectives, the study will also describe molecular profile, cytogenetic risk, clinical outcomes, and healthcare resource utilization of treated B-cell ALL R/R and AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old at diagnosis
* Confirmed diagnosis of relapsed/refractory B-cell ALL or de novo AML diagnosed between 01 January 2015 and 31 December 2019
* At least 1 line of treatment for R/R B-cell ALL or de novo AML within the study period

Exclusion Criteria:

* Patients with no medical chart available
* Patients with unreliable data as per investigator's opinion (e.g. excessive missing data or inconsistence data)
* Patients that have participated in any interventional clinical trial for relapsed/refractory B-cell ALL or AML at any moment
* Patients with secondary AML
* Patients with any concomitant primary malignancy
* Patients with acute promyelocytic leukemia (APL)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old at diagnosis, with de novo AML or R/R B-cell ALL diagnosed between 01 January 2015 and 31 December 2019, as documented in the medical chart and according to the physician's notes, and with at least 1 line of treatment for AML or R/R ALL within the study period.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Argentina (5):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - FUNDALEU - Fundacion para combatir la Leucemia, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
  - Sanatorio Allende, Córdoba
- Brazil (6):
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Fundação Doutor Amaral Carvalho, Jaú, SAO Paulo / Brazil
  - Instituto COI de Pesquisa, Rio de Janeiro
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
  - Hospital Beneficência Portuguesa de São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Hospital Guillermo Grant Benavente, Concepción, Chile
- Colombia (2):
  - Fundacion Santa Fe de Bogota, Bogotá
  - Oncomedica SA, Montería

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed acute myeloid leukemia (AML) or with relapsed/refractory (R/R) B-cell acute lymphoblastic leukemia (ALL) diagnosed between 01-Jan-2015 and 31-Dec-2019 were included in the study. Data was extracted from participants medical charts and was analyzed retrospectively over approximately 11 months.
Pre-assignment Details: A total of 628 participants were screened of which 39 did not meet eligibility criteria and were excluded and 589 participants were included in the study.
Groups:
- Newly AML: Participants newly diagnosed with AML between 01-Jan-2015 and 31-Dec-2019 and who received at least one line of treatment for AML were included.
- R/R B-cell ALL: Participants with a confirmed diagnosis of R/R B cell ALL between 01-Jan-2015 and 31-Dec-2019 and who received at least one line of treatment for R/R B-cell ALL were included.
Period: Overall Study
Arm/Group | Newly AML | R/R B-cell ALL
Started | 518 | 71
Completed | 518 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly AML | R/R B-cell ALL | Total
Number analyzed (Participants) | 518 | 71 | 589
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (16.7) | 36.6 (15.5) | 52.5 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 31 | 295
  Male | 254 | 40 | 294
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the baseline measure.
  Participants
    number analyzed (Participants) | 493 | 66 | 559
    American Indian | 38 | 9 | 47
    Asian | 2 | 0 | 2
    Black or African American | 21 | 4 | 25
    White or Caucasian | 363 | 33 | 396
    Other | 69 | 20 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Health Insurance Type
Description: Number of participants according to type of health insurance (public or private) were reported in this outcome measure.
Time Frame: At index (anytime between 01-Jan-2015 and 31-Dec-2019; approximately 5 years); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants
  Private | 265 | 44
  Public | 253 | 27

2. Primary Outcome: Number of Participants According to Country of Residence
Description: Number of participants according to country of residence such as Argentina, Brazil, Chile, and Colombia were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants
  Argentina | 166 | 23
  Brazil | 205 | 27
  Chile | 63 | 0
  Colombia | 84 | 21

3. Primary Outcome: Number of Participants With Comorbidities
Description: Number of participants with any comorbidity at de novo AML or B-cell ALL diagnosis were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants | 273 | 23

4. Primary Outcome: Number of Participants According to Family History of Hematological Malignancies
Description: Number of participants who had a family history of hematological malignancies were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants | 21 | 3

5. Primary Outcome: Number of Participants With Prior Exposure to Toxic Agents
Description: Number of participants who had any prior exposure to toxic agents were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants | 11 | 3

6. Primary Outcome: Number of Participants With Prior Exposure to a High Dose of Radiation
Description: Number of participants with prior exposure to a high dose of radiation were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants | 2 | 1

7. Primary Outcome: Number of Participants According to Reason for Exposure to High Dose of Radiation
Description: Number of participants according to reason for exposure to high dose of radiation were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 2 | 1
Participants
  Therapeutic radiation for other cancers | 2 | 0
  Accidental exposures | 0 | 0
  Other | 0 | 1

8. Primary Outcome: Number of Participants With Bleeding History
Description: Number of participants with bleeding history were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants | 30 | 6

9. Primary Outcome: Number of Participants With Tobacco Consumption Habits
Description: Participants with tobacco consumption habits (i.e., Non-smoker, Ex-smoker and others) were reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 479 | 70
Participants
  Non-smoker | 343 | 55
  Ex-smoker | 85 | 10
  Other | 51 | 5

10. Primary Outcome: Number of Participants According to Eastern Cooperative Oncology Group (ECOG) Performance Status Scores
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. In this outcome measure, data for ECOG status (0, 1, 2, 3 and 4) was reported.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study., Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 387 | 57
Participants
  0 | 136 | 29
  1 | 185 | 21
  2 | 45 | 7
  3 | 16 | 0
  4 | 5 | 0

11. Primary Outcome: Number of Participants According to Karnofsky Performance Scores
Description: Karnofsky performance score was used to quantify participant's general well-being and activities of daily life and participants were classified based on their functional impairment. Karnofsky performance score was 11 level score which ranges between 0 (death) to 100 (no evidence of disease). Score:100=normal no complaints; no disease evidence,90=able to carry normal activity; minor signs/symptoms of disease,80=normal activity with effort; some signs/symptoms, 70=cares for self; unable to carry normal activity, 60=required occasional assistance, able to care for personal needs, 50=required considerable assistance & frequent medical care, 40=disabled; required special care/assistance,30=severely disabled; hospital admission indicated;20=very sick; hospital admission necessary,10=moribund and 0=dead.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 337 | 50
Participants
  100 | 110 | 27
  90 | 107 | 12
  80 | 69 | 7
  70 | 29 | 2
  60 | 4 | 2
  50 | 14 | 0
  40 | 4 | 0
  30 | 0 | 0
  20 | 0 | 0
  10 | 0 | 0

12. Primary Outcome: Number of Participants According to Year of Diagnosis
Description: Number of participants according to the year of diagnosis for newly AML or R/R B-cell ALL were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Participants
  2015 | 88 | 13
  2016 | 102 | 15
  2017 | 103 | 4
  2018 | 125 | 21
  2019 | 100 | 18

13. Primary Outcome: Number of Participants According to Classification for Standard Newly AML Therapy
Description: Number of participants classified as fit or unfit for the standard newly AML therapy according to different lines of treatment (LOT) were reported in this outcome measure.
Time Frame: From diagnosis until loss of follow-up or death (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. and 'Number Analyzed' signifies participants evaluable for the specified rows. Only newly AML participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 489
Participants
  LOT1: Fit | 390
  LOT1: Unfit | 99
  LOT2: number analyzed (Participants) | 260
  LOT2: Fit | 217
  LOT2: Unfit | 43
  LOT3: number analyzed (Participants) | 134
  LOT3: Fit | 102
  LOT3: Unfit | 32
  LOT4: number analyzed (Participants) | 53
  LOT4: Fit | 40
  LOT4: Unfit | 13
  LOT5-LOT7: number analyzed (Participants) | 25
  LOT5-LOT7: Fit | 15
  LOT5-LOT7: Unfit | 10

14. Primary Outcome: Number of Participants According to Drug Regimen Prescribed for Newly AML
Description: A regimen was defined as a plan for the dose, schedule, and length of treatment. A regimen could be a treatment that consisted of one or combined (two or more) drugs. Number of participants according to drug regimen prescribed for newly AML were reported by each line of treatment (LOT). Drug regimen included standard 7+3, Histone deacetylases (HDACs), Low-dose Cytarabine (LDAC), FLAG (fludarabine + high-dose cytarabine + G-CSF (Granulocyte colony-stimulating factor), FLAG-IDA Regimen (Fludarabine, Cytarabine, Idarubicin and G-CSF), Hypomethylating agents (HMA), CLAG (Cladribine + Cytarabine + G-CSF), MEC (mitoxantrone, etoposide and intermediate dose cytarabine), MICE and other.
Time Frame: as for outcome 13
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows. Only newly AML participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 518
Participants
  Standard 7+3 (LOT1) | 390
  HDAC (LOT1) | 3
  LDAC (LOT1) | 25
  FLAG (LOT1) | 3
  FLAG-IDA (LOT1) | 3
  HMA (LOT1) | 47
  CLAG (LOT1) | 0
  MEC (LOT1) | 0
  MICE (LOT1) | 0
  Other (LOT1) | 47
  Standard 7+3 (LOT2): number analyzed (Participants) | 276
  Standard 7+3 (LOT2) | 9
  HDAC (LOT2): number analyzed (Participants) | 276
  HDAC (LOT2) | 85
  LDAC (LOT2): number analyzed (Participants) | 276
  LDAC (LOT2) | 7
  FLAG (LOT2): number analyzed (Participants) | 276
  FLAG (LOT2) | 3
  FLAG-IDA (LOT2): number analyzed (Participants) | 276
  FLAG-IDA (LOT2) | 66
  HMA (LOT2): number analyzed (Participants) | 276
  HMA (LOT2) | 26
  CLAG (LOT2): number analyzed (Participants) | 276
  CLAG (LOT2) | 0
  MEC (LOT2): number analyzed (Participants) | 276
  MEC (LOT2) | 24
  MICE (LOT2): number analyzed (Participants) | 276
  MICE (LOT2) | 0
  Other (LOT2): number analyzed (Participants) | 276
  Other (LOT2) | 56
  Standard 7+3 (LOT3): number analyzed (Participants) | 144
  Standard 7+3 (LOT3) | 3
  HDAC (LOT3): number analyzed (Participants) | 144
  HDAC (LOT3) | 24
  LDAC (LOT3): number analyzed (Participants) | 144
  LDAC (LOT3) | 5
  FLAG (LOT3): number analyzed (Participants) | 144
  FLAG (LOT3) | 5
  FLAG-IDA (LOT3): number analyzed (Participants) | 144
  FLAG-IDA (LOT3) | 36
  HMA (LOT3): number analyzed (Participants) | 144
  HMA (LOT3) | 30
  CLAG (LOT3): number analyzed (Participants) | 144
  CLAG (LOT3) | 1
  MEC (LOT3): number analyzed (Participants) | 144
  MEC (LOT3) | 9
  MICE (LOT3): number analyzed (Participants) | 144
  MICE (LOT3) | 0
  Other (LOT3): number analyzed (Participants) | 144
  Other (LOT3) | 31
  Standard 7+3 (LOT4): number analyzed (Participants) | 60
  Standard 7+3 (LOT4) | 3
  HDAC (LOT4): number analyzed (Participants) | 60
  HDAC (LOT4) | 20
  LDAC (LOT4): number analyzed (Participants) | 60
  LDAC (LOT4) | 1
  FLAG (LOT4): number analyzed (Participants) | 60
  FLAG (LOT4) | 0
  FLAG-IDA (LOT4): number analyzed (Participants) | 60
  FLAG-IDA (LOT4) | 3
  HMA (LOT4): number analyzed (Participants) | 60
  HMA (LOT4) | 13
  CLAG (LOT4): number analyzed (Participants) | 60
  CLAG (LOT4) | 1
  MEC (LOT4): number analyzed (Participants) | 60
  MEC (LOT4) | 5
  MICE (LOT4): number analyzed (Participants) | 60
  MICE (LOT4) | 0
  Other (LOT4): number analyzed (Participants) | 60
  Other (LOT4) | 14
  Standard 7+3 (LOT5-LOT7): number analyzed (Participants) | 28
  Standard 7+3 (LOT5-LOT7) | 2
  HDAC (LOT5-LOT7): number analyzed (Participants) | 28
  HDAC (LOT5-LOT7) | 2
  LDAC (LOT5-LOT7): number analyzed (Participants) | 28
  LDAC (LOT5-LOT7) | 0
  FLAG (LOT5-LOT7): number analyzed (Participants) | 28
  FLAG (LOT5-LOT7) | 0
  FLAG-IDA (LOT5-LOT7): number analyzed (Participants) | 28
  FLAG-IDA (LOT5-LOT7) | 7
  HMA (LOT5-LOT7): number analyzed (Participants) | 28
  HMA (LOT5-LOT7) | 4
  CLAG (LOT5-LOT7): number analyzed (Participants) | 28
  CLAG (LOT5-LOT7) | 0
  MEC (LOT5-LOT7): number analyzed (Participants) | 28
  MEC (LOT5-LOT7) | 3
  MICE (LOT5-LOT7): number analyzed (Participants) | 28
  MICE (LOT5-LOT7) | 0
  Other (LOT5-LOT7): number analyzed (Participants) | 28
  Other (LOT5-LOT7) | 10

15. Primary Outcome: Number of Participants According to Drug Regimen Prescribed for R/R B-cell ALL
Description: A regimen was defined as a plan for the dose, schedule, and length of treatment. A regimen could be a treatment that consisted of one or combined (two or more) drugs. Number of participants according to drug regimen prescribed for R/R B-cell ALL were reported by each LOT is reported. Drug regimen included Hyper- CVAD (hyperfractionated cyclophosphamide, vincristine, doxorubicin, and prednisolone), German multicenter study group for ALL (GMALL), Group for Research on Adult Acute Lymphoblastic Leukemia (GRAAL), Berlin-Frankfurt-Münster (BFM), Inotuzumab, Blinatumomab, Chimeric antigen receptor T-cell therapies (CAR-T), Tyrosine kinase inhibitors (TKI), FLAG (fludarabine + high-dose cytarabine + G-CSF), FLAG-IDA Regimen (Fludarabine, Cytarabine, Idarubicin and G-CSF), Other. One participant could be prescribed more than 1 drug regimen.
Time Frame: as for outcome 13
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows. Only R/R B-cell ALL participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 71
Participants
  Hyper-CVAD (LOT1) | 16
  GMALL (LOT1) | 0
  GRAAL (LOT1) | 11
  BFM (LOT1) | 15
  Inotuzumab (LOT1) | 0
  Blinatumomab (LOT1) | 0
  Car T-cell (LOT1) | 0
  TKI inhibitor (LOT1) | 4
  FLAG (LOT1) | 2
  FLAG-IDA (LOT1) | 1
  Other (LOT1) | 29
  Hyper-CVAD (LOT2): number analyzed (Participants) | 53
  Hyper-CVAD (LOT2) | 14
  GMALL (LOT2): number analyzed (Participants) | 53
  GMALL (LOT2) | 0
  GRAAL (LOT2): number analyzed (Participants) | 53
  GRAAL (LOT2) | 1
  BFM (LOT2): number analyzed (Participants) | 53
  BFM (LOT2) | 2
  Inotuzumab (LOT2): number analyzed (Participants) | 53
  Inotuzumab (LOT2) | 0
  Blinatumomab (LOT2): number analyzed (Participants) | 53
  Blinatumomab (LOT2) | 1
  Car T-cell (LOT2): number analyzed (Participants) | 53
  Car T-cell (LOT2) | 0
  TKI inhibitor (LOT2): number analyzed (Participants) | 53
  TKI inhibitor (LOT2) | 2
  FLAG (LOT2): number analyzed (Participants) | 53
  FLAG (LOT2) | 1
  FLAG-IDA (LOT2): number analyzed (Participants) | 53
  FLAG-IDA (LOT2) | 15
  Other (LOT2): number analyzed (Participants) | 53
  Other (LOT2) | 22
  Hyper-CVAD (LOT3): number analyzed (Participants) | 26
  Hyper-CVAD (LOT3) | 3
  GMALL (LOT3): number analyzed (Participants) | 26
  GMALL (LOT3) | 0
  GRAAL (LOT3): number analyzed (Participants) | 26
  GRAAL (LOT3) | 0
  BFM (LOT3): number analyzed (Participants) | 26
  BFM (LOT3) | 1
  Inotuzumab (LOT3): number analyzed (Participants) | 26
  Inotuzumab (LOT3) | 0
  Blinatumomab (LOT3): number analyzed (Participants) | 26
  Blinatumomab (LOT3) | 5
  Car T-cell (LOT3): number analyzed (Participants) | 26
  Car T-cell (LOT3) | 0
  TKI inhibitor (LOT3): number analyzed (Participants) | 26
  TKI inhibitor (LOT3) | 2
  FLAG (LOT3): number analyzed (Participants) | 26
  FLAG (LOT3) | 0
  FLAG-IDA (LOT3): number analyzed (Participants) | 26
  FLAG-IDA (LOT3) | 5
  Other (LOT3): number analyzed (Participants) | 26
  Other (LOT3) | 12
  Hyper-CVAD (LOT4): number analyzed (Participants) | 12
  Hyper-CVAD (LOT4) | 2
  GMALL (LOT4): number analyzed (Participants) | 12
  GMALL (LOT4) | 0
  GRAAL (LOT4): number analyzed (Participants) | 12
  GRAAL (LOT4) | 0
  BFM (LOT4): number analyzed (Participants) | 12
  BFM (LOT4) | 0
  Inotuzumab (LOT4): number analyzed (Participants) | 12
  Inotuzumab (LOT4) | 1
  Blinatumomab (LOT4): number analyzed (Participants) | 12
  Blinatumomab (LOT4) | 1
  Car T-cell (LOT4): number analyzed (Participants) | 12
  Car T-cell (LOT4) | 0
  TKI inhibitor (LOT4): number analyzed (Participants) | 12
  TKI inhibitor (LOT4) | 2
  FLAG (LOT4): number analyzed (Participants) | 12
  FLAG (LOT4) | 0
  FLAG-IDA (LOT4): number analyzed (Participants) | 12
  FLAG-IDA (LOT4) | 3
  Other (LOT4): number analyzed (Participants) | 12
  Other (LOT4) | 7
  Hyper-CVAD (LOT5-LOT7): number analyzed (Participants) | 5
  Hyper-CVAD (LOT5-LOT7) | 0
  GMALL (LOT5-LOT7): number analyzed (Participants) | 5
  GMALL (LOT5-LOT7) | 0
  GRAAL (LOT5-LOT7): number analyzed (Participants) | 5
  GRAAL (LOT5-LOT7) | 0
  BFM (LOT5-LOT7): number analyzed (Participants) | 5
  BFM (LOT5-LOT7) | 0
  Inotuzumab (LOT5-LOT7): number analyzed (Participants) | 5
  Inotuzumab (LOT5-LOT7) | 2
  Blinatumomab (LOT5-LOT7): number analyzed (Participants) | 5
  Blinatumomab (LOT5-LOT7) | 1
  Car T-cell (LOT5-LOT7): number analyzed (Participants) | 5
  Car T-cell (LOT5-LOT7) | 0
  TKI inhibitor (LOT5-LOT7): number analyzed (Participants) | 5
  TKI inhibitor (LOT5-LOT7) | 0
  FLAG (LOT5-LOT7): number analyzed (Participants) | 5
  FLAG (LOT5-LOT7) | 0
  FLAG-IDA (LOT5-LOT7): number analyzed (Participants) | 5
  FLAG-IDA (LOT5-LOT7) | 0
  Other (LOT5-LOT7): number analyzed (Participants) | 5
  Other (LOT5-LOT7) | 4

16. Primary Outcome: Number of Participants Prescribed Gemtuzumab, Midostaurin or Venetoclax Treatment in Newly AML
Description: Number of participants prescribed Gemtuzumab, Midostaurin or Venetoclax treatment in newly AML according to different LOT were reported in this outcome measure.
Time Frame: as for outcome 13
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for the specified rows. Only newly AML participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 41
Participants
  Gemtuzumab (LOT1): number analyzed (Participants) | 11
  Gemtuzumab (LOT1) | 0
  Midostaurin (LOT1): number analyzed (Participants) | 11
  Midostaurin (LOT1) | 10
  Venetoclax (LOT1): number analyzed (Participants) | 11
  Venetoclax (LOT1) | 1
  Gemtuzumab (LOT2): number analyzed (Participants) | 12
  Gemtuzumab (LOT2) | 1
  Midostaurin (LOT2): number analyzed (Participants) | 12
  Midostaurin (LOT2) | 9
  Venetoclax (LOT2): number analyzed (Participants) | 12
  Venetoclax (LOT2) | 3
  Gemtuzumab (LOT3): number analyzed (Participants) | 12
  Gemtuzumab (LOT3) | 2
  Midostaurin (LOT3): number analyzed (Participants) | 12
  Midostaurin (LOT3) | 3
  Venetoclax (LOT3): number analyzed (Participants) | 12
  Venetoclax (LOT3) | 7
  Gemtuzumab (LOT4): number analyzed (Participants) | 3
  Gemtuzumab (LOT4) | 0
  Midostaurin (LOT4): number analyzed (Participants) | 3
  Midostaurin (LOT4) | 1
  Venetoclax (LOT4): number analyzed (Participants) | 3
  Venetoclax (LOT4) | 2
  Gemtuzumab (LOT5-LOT7): number analyzed (Participants) | 3
  Gemtuzumab (LOT5-LOT7) | 0
  Midostaurin (LOT5-LOT7): number analyzed (Participants) | 3
  Midostaurin (LOT5-LOT7) | 0
  Venetoclax (LOT5-LOT7): number analyzed (Participants) | 3
  Venetoclax (LOT5-LOT7) | 3

17. Primary Outcome: Number of Participants According to Regimen Type in Newly AML
Description: Number of participants according to drug regimen prescribed for newly AML is reported by each LOT. Induction was the first phase of treatment. Consolidation was given after the participant had recovered from induction. Maintenance was given to maintain the remission and further prevent a relapse. Salvage was used when a disease did not respond to all other standard treatments tried.
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 515
Participants
  Induction (LOT1) | 458
  Consolidation (LOT1) | 92
  Maintenance (LOT1) | 7
  Salvage (LOT1) | 2
  Other (LOT1) | 55
  Induction (LOT2): number analyzed (Participants) | 277
  Induction (LOT2) | 46
  Consolidation (LOT2): number analyzed (Participants) | 277
  Consolidation (LOT2) | 126
  Maintenance (LOT2): number analyzed (Participants) | 277
  Maintenance (LOT2) | 7
  Salvage (LOT2): number analyzed (Participants) | 277
  Salvage (LOT2) | 93
  Other (LOT2): number analyzed (Participants) | 277
  Other (LOT2) | 27
  Induction (LOT3): number analyzed (Participants) | 145
  Induction (LOT3) | 11
  Consolidation (LOT3): number analyzed (Participants) | 145
  Consolidation (LOT3) | 42
  Maintenance (LOT3): number analyzed (Participants) | 145
  Maintenance (LOT3) | 10
  Salvage (LOT3): number analyzed (Participants) | 145
  Salvage (LOT3) | 73
  Other (LOT3): number analyzed (Participants) | 145
  Other (LOT3) | 17
  Induction (LOT4): number analyzed (Participants) | 60
  Induction (LOT4) | 3
  Consolidation (LOT4): number analyzed (Participants) | 60
  Consolidation (LOT4) | 27
  Maintenance (LOT4): number analyzed (Participants) | 60
  Maintenance (LOT4) | 5
  Salvage (LOT4): number analyzed (Participants) | 60
  Salvage (LOT4) | 22
  Other (LOT4): number analyzed (Participants) | 60
  Other (LOT4) | 6
  Induction (LOT5-LOT7): number analyzed (Participants) | 28
  Induction (LOT5-LOT7) | 1
  Consolidation (LOT5-LOT7): number analyzed (Participants) | 28
  Consolidation (LOT5-LOT7) | 3
  Maintenance (LOT5-LOT7): number analyzed (Participants) | 28
  Maintenance (LOT5-LOT7) | 4
  Salvage (LOT5-LOT7): number analyzed (Participants) | 28
  Salvage (LOT5-LOT7) | 16
  Other (LOT5-LOT7): number analyzed (Participants) | 28
  Other (LOT5-LOT7) | 5

18. Primary Outcome: Treatment Duration
Description: The duration of treatment according to different treatment lines were reported.
Time Frame: From start of treatment until end of treatment, disease progression, death or loss of follow-up (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 503 | 67
Months
  LOT1 | 2.1 (4.0) | 6.4 (7.9)
  LOT2: number analyzed (Participants) | 270 | 53
  LOT2 | 2.2 (3.3) | 3.9 (7.1)
  LOT3: number analyzed (Participants) | 140 | 26
  LOT3 | 2.3 (4.2) | 1.7 (2.0)
  LOT4: number analyzed (Participants) | 57 | 12
  LOT4 | 1.8 (2.5) | 6.0 (18.2)
  LOT5-LOT7: number analyzed (Participants) | 27 | 6
  LOT5-LOT7 | 2.2 (4.2) | 2.6 (3.7)

19. Primary Outcome: Time to Next Treatment
Description: Time to next treatment was considered as the time from the start date of the front-line therapy to the start date of a subsequent line of therapy. Participants without a subsequent line of therapy were censored at study enrollment, last visit, last contact, or death, whichever comes first.
Time Frame: From start of front-line therapy until start of subsequent line of therapy, last visit/contact/death (up to maximum of 94.6 months);data collected and observed retrospectively over 11 month
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 275 | 53
Months
  LOT1 to LOT2 | 1.6 [1.5 to 1.7] | 8.4 [6.1 to 14.5]
  LOT2 to LOT3: number analyzed (Participants) | 143 | 26
  LOT2 to LOT3 | 2.9 [2.2 to 4.8] | 2.6 [1.8 to 13.5]
  LOT3 to LOT4: number analyzed (Participants) | 58 | 12
  LOT3 to LOT4 | 2.0 [1.5 to 2.6] | 2.4 [1.8 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.
  LOT4 to LOT5: number analyzed (Participants) | 22 | 3
  LOT4 to LOT5 | 4.2 [3.0 to 8.2] | 2.7 [2.1 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.
  LOT5 to LOT6, LOT6 to LOT7: number analyzed (Participants) | 6 | 3
  LOT5 to LOT6, LOT6 to LOT7 | 4.8 [4.2 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.9 [2.5 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

20. Primary Outcome: Total Number of Cycles
Description: Total number of cycles according to each line of treatment is reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 486 | 64
Cycles
  LOT1 | 2.2 (3.1) | 3.1 (2.5)
  LOT2: number analyzed (Participants) | 271 | 50
  LOT2 | 2.2 (2.6) | 2.7 (4.0)
  LOT3: number analyzed (Participants) | 134 | 24
  LOT3 | 2.2 (3.0) | 2.6 (2.0)
  LOT4: number analyzed (Participants) | 56 | 12
  LOT4 | 2.0 (2.1) | 6.5 (16.9)
  LOT5-LOT7: number analyzed (Participants) | 24 | 5
  LOT5-LOT7 | 2.0 (1.9) | 1.4 (0.5)

21. Primary Outcome: Number of Participants Who Withdrew Regimen
Description: Number of participants who withdrew regimen according to each line of treatment is reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 502 | 70
Participants
  LOT1 | 86 | 8
  LOT2: number analyzed (Participants) | 271 | 52
  LOT2 | 35 | 12
  LOT3: number analyzed (Participants) | 139 | 26
  LOT3 | 19 | 10
  LOT4: number analyzed (Participants) | 58 | 12
  LOT4 | 8 | 5
  LOT5-LOT7: number analyzed (Participants) | 26 | 5
  LOT5-LOT7 | 2 | 1

22. Primary Outcome: Number of Participants According to Reasons for Withdrawing Regimen
Description: Number of participants according to reasons such as progression of the disease, Adverse event toxicity, participants refusal to continue the treatment scheme, cost related or access barriers and other for withdrawing regimen according to each line of treatment were reported in this outcome measure. One participant could have more than one reason for withdrawing regimen.
Time Frame: as for outcome 18
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants with reasons available for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 86 | 12
Participants
  Progression of the disease (LOT1): number analyzed (Participants) | 86 | 8
  Progression of the disease (LOT1) | 14 | 3
  Adverse event-toxicity (LOT1): number analyzed (Participants) | 86 | 8
  Adverse event-toxicity (LOT1) | 28 | 2
  Participant's refusal to continue the treatment scheme (LOT1): number analyzed (Participants) | 86 | 8
  Participant's refusal to continue the treatment scheme (LOT1) | 0 | 0
  Cost-related or access barriers (LOT1): number analyzed (Participants) | 86 | 8
  Cost-related or access barriers (LOT1) | 0 | 0
  Other (LOT1): number analyzed (Participants) | 86 | 8
  Other (LOT1) | 44 | 3
  Progression of the disease (LOT2): number analyzed (Participants) | 35 | 12
  Progression of the disease (LOT2) | 11 | 3
  Adverse event-toxicity (LOT2): number analyzed (Participants) | 35 | 12
  Adverse event-toxicity (LOT2) | 9 | 4
  Participant's refusal to continue the treatment scheme (LOT2): number analyzed (Participants) | 35 | 12
  Participant's refusal to continue the treatment scheme (LOT2) | 1 | 0
  Cost-related or access barriers (LOT2): number analyzed (Participants) | 35 | 12
  Cost-related or access barriers (LOT2) | 0 | 0
  Other (LOT2): number analyzed (Participants) | 35 | 12
  Other (LOT2) | 15 | 5
  Progression of the disease (LOT3): number analyzed (Participants) | 19 | 10
  Progression of the disease (LOT3) | 5 | 4
  Adverse event-toxicity (LOT3): number analyzed (Participants) | 19 | 10
  Adverse event-toxicity (LOT3) | 4 | 1
  Participant's refusal to continue the treatment scheme (LOT3): number analyzed (Participants) | 19 | 10
  Participant's refusal to continue the treatment scheme (LOT3) | 0 | 0
  Cost-related or access barriers (LOT3): number analyzed (Participants) | 19 | 10
  Cost-related or access barriers (LOT3) | 1 | 0
  Other (LOT3): number analyzed (Participants) | 19 | 10
  Other (LOT3) | 9 | 5
  Progression of the disease (LOT4): number analyzed (Participants) | 8 | 4
  Progression of the disease (LOT4) | 4 | 0
  Adverse event-toxicity (LOT4): number analyzed (Participants) | 8 | 4
  Adverse event-toxicity (LOT4) | 1 | 2
  Participant's refusal to continue the treatment scheme (LOT4): number analyzed (Participants) | 8 | 4
  Participant's refusal to continue the treatment scheme (LOT4) | 0 | 0
  Cost-related or access barriers (LOT4): number analyzed (Participants) | 8 | 4
  Cost-related or access barriers (LOT4) | 0 | 0
  Other (LOT4): number analyzed (Participants) | 8 | 4
  Other (LOT4) | 3 | 2
  Progression of the disease (LOT5-LOT7): number analyzed (Participants) | 2 | 1
  Progression of the disease (LOT5-LOT7) | 2 | 0
  Adverse event-toxicity (LOT5-LOT7): number analyzed (Participants) | 2 | 1
  Adverse event-toxicity (LOT5-LOT7) | 0 | 0
  Participant's refusal to continue the treatment scheme (LOT5-LOT7): number analyzed (Participants) | 2 | 1
  Participant's refusal to continue the treatment scheme (LOT5-LOT7) | 0 | 0
  Cost-related or access barriers (LOT5-LOT7): number analyzed (Participants) | 2 | 1
  Cost-related or access barriers (LOT5-LOT7) | 0 | 0
  Other (LOT5-LOT7): number analyzed (Participants) | 2 | 1
  Other (LOT5-LOT7) | 0 | 1

23. Primary Outcome: Number of Participants With Dose Reduction
Description: Number of participants with dose reduction according to each line of treatment were reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 487 | 67
Participants
  LOT1 | 84 | 9
  LOT2: number analyzed (Participants) | 269 | 51
  LOT2 | 37 | 7
  LOT3: number analyzed (Participants) | 136 | 25
  LOT3 | 15 | 2
  LOT4: number analyzed (Participants) | 56 | 12
  LOT4 | 3 | 1
  LOT5-LOT7: number analyzed (Participants) | 24 | 5
  LOT5-LOT7 | 1 | 1

24. Primary Outcome: Number of Participants With Central Nervous System (CNS) Involvement at Disease Progression
Description: Number of participants with CNS involvement at disease progression according to each line of treatment were reported in this outcome measure.
Time Frame: At disease progression (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 33 | 9
Participants
  LOT1 | 1 | 0
  LOT2: number analyzed (Participants) | 19 | 5
  LOT2 | 1 | 1
  LOT3: number analyzed (Participants) | 9 | 3
  LOT3 | 2 | 2
  LOT4: number analyzed (Participants) | 6 | 0
  LOT4 | 1 | 0
  LOT5-LOT7: number analyzed (Participants) | 2 | 0
  LOT5-LOT7 | 0 | 0

25. Primary Outcome: Duration of Radiotherapy
Description: Mean duration of radiotherapy according to each line of treatment is reported in this outcome measure.
Time Frame: as for outcome 18
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 2 | 3
Months
  LOT1: number analyzed (Participants) | 1 | 3
  LOT1 | 0.3 (0) | 0.7 (0.6)
  LOT2: number analyzed (Participants) | 0 | 0
  LOT3: number analyzed (Participants) | 1 | 0
  LOT3 | 0.5 |
  LOT4: number analyzed (Participants) | 0 | 0
  LOT5-LOT7: number analyzed (Participants) | 0 | 0

26. Primary Outcome: Dose of Radiotherapy
Description: Mean dose of radiotherapy according to each line of treatment is reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Rad
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 3 | 3
Rad
  LOT1: number analyzed (Participants) | 1 | 3
  LOT1 | 300 (NA) — Standard deviation could not be calculated as only one participants was analyzed. | 2267 (1553)
  LOT2: number analyzed (Participants) | 1 | 0
  LOT2 | 25 (NA) — Standard deviation could not be calculated as only one participants was analyzed. |
  LOT3: number analyzed (Participants) | 1 | 1
  LOT3 | 2400 (NA) — Standard deviation could not be calculated as only one participants was analyzed. | 24
  LOT4: number analyzed (Participants) | 0 | 0
  LOT5-LOT7: number analyzed (Participants) | 0 | 0

27. Primary Outcome: Number of Participants According to Location of Application of Radiotherapy
Description: Number of participants according to location of application of radiotherapy according to each line of treatment is reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 2 | 3
Participants
  LOT1: number analyzed (Participants) | 1 | 3
  LOT1: CNS (cranial irradiation) | 0 | 2
  LOT1: Total body irradiation | 0 | 0
  LOT1: Other | 1 | 1
  LOT2: number analyzed (Participants) | 2 | 0
  LOT2: CNS (cranial irradiation) | 1 | 0
  LOT2: Total body irradiation | 1 | 0
  LOT2: Other | 0 | 0
  LOT3: number analyzed (Participants) | 1 | 2
  LOT3: CNS (cranial irradiation) | 0 | 1
  LOT3: Total body irradiation | 0 | 1
  LOT3: Other | 1 | 0
  LOT4: number analyzed (Participants) | 0 | 0
  LOT4: CNS (cranial irradiation) | 0 | 0
  LOT4: Total body irradiation | 0 | 0
  LOT4: Other | 0 | 0
  LOT5-LOT7: number analyzed (Participants) | 0 | 0
  LOT5-LOT7: CNS (cranial irradiation) | 0 | 0
  LOT5-LOT7: Total body irradiation | 0 | 0
  LOT5-LOT7: Other | 0 | 0

28. Primary Outcome: Number of Participants According to Intrathecal Chemotherapy
Description: Number of participants according to intrathecal chemotherapy such as methotrexate, cytarabine, prednisone, dexamethasone, other according to each line of treatment is reported in this outcome measure. One participant may receive more than one intrathecal chemotherapy.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 509 | 69
Participants
  Intrathecal chemotherapy (LOT1) | 75 | 49
  Methotrexate (LOT1): number analyzed (Participants) | 75 | 49
  Methotrexate (LOT1) | 42 | 46
  Cytarabine (LOT1): number analyzed (Participants) | 75 | 49
  Cytarabine (LOT1) | 74 | 44
  Prednisone (LOT1): number analyzed (Participants) | 75 | 49
  Prednisone (LOT1) | 0 | 1
  Dexamethasone (LOT1): number analyzed (Participants) | 75 | 49
  Dexamethasone (LOT1) | 70 | 41
  Other (LOT1): number analyzed (Participants) | 75 | 49
  Other (LOT1) | 5 | 0
  Intrathecal chemotherapy (LOT2): number analyzed (Participants) | 270 | 52
  Intrathecal chemotherapy (LOT2) | 35 | 29
  Methotrexate (LOT2): number analyzed (Participants) | 35 | 29
  Methotrexate (LOT2) | 18 | 28
  Cytarabine (LOT2): number analyzed (Participants) | 35 | 29
  Cytarabine (LOT2) | 33 | 24
  Prednisone (LOT2): number analyzed (Participants) | 35 | 29
  Prednisone (LOT2) | 0 | 0
  Dexamethasone (LOT2): number analyzed (Participants) | 35 | 29
  Dexamethasone (LOT2) | 32 | 25
  Other (LOT2): number analyzed (Participants) | 35 | 29
  Other (LOT2) | 4 | 1
  Intrathecal chemotherapy (LOT3): number analyzed (Participants) | 140 | 25
  Intrathecal chemotherapy (LOT3) | 10 | 10
  Methotrexate (LOT3): number analyzed (Participants) | 10 | 10
  Methotrexate (LOT3) | 6 | 10
  Cytarabine (LOT3): number analyzed (Participants) | 10 | 10
  Cytarabine (LOT3) | 9 | 8
  Prednisone (LOT3): number analyzed (Participants) | 10 | 10
  Prednisone (LOT3) | 0 | 0
  Dexamethasone (LOT3): number analyzed (Participants) | 10 | 10
  Dexamethasone (LOT3) | 8 | 9
  Other (LOT3): number analyzed (Participants) | 10 | 10
  Other (LOT3) | 1 | 0
  Intrathecal chemotherapy (LOT4): number analyzed (Participants) | 59 | 11
  Intrathecal chemotherapy (LOT4) | 6 | 5
  Methotrexate (LOT4): number analyzed (Participants) | 6 | 5
  Methotrexate (LOT4) | 5 | 4
  Cytarabine (LOT4): number analyzed (Participants) | 6 | 5
  Cytarabine (LOT4) | 6 | 5
  Prednisone (LOT4): number analyzed (Participants) | 6 | 5
  Prednisone (LOT4) | 0 | 0
  Dexamethasone (LOT4): number analyzed (Participants) | 6 | 5
  Dexamethasone (LOT4) | 2 | 5
  Other (LOT4): number analyzed (Participants) | 6 | 5
  Other (LOT4) | 2 | 0
  Intrathecal chemotherapy (LOT5-LOT7): number analyzed (Participants) | 28 | 5
  Intrathecal chemotherapy (LOT5-LOT7) | 3 | 2
  Methotrexate (LOT5-LOT7): number analyzed (Participants) | 3 | 2
  Methotrexate (LOT5-LOT7) | 2 | 2
  Cytarabine (LOT5-LOT7): number analyzed (Participants) | 3 | 2
  Cytarabine (LOT5-LOT7) | 3 | 2
  Prednisone (LOT5-LOT7): number analyzed (Participants) | 3 | 2
  Prednisone (LOT5-LOT7) | 0 | 0
  Dexamethasone (LOT5-LOT7): number analyzed (Participants) | 3 | 2
  Dexamethasone (LOT5-LOT7) | 2 | 2
  Other (LOT5-LOT7): number analyzed (Participants) | 3 | 2
  Other (LOT5-LOT7) | 1 | 0

29. Primary Outcome: Number of Participants With Stem Cell Transplant (SCT)
Description: Number of participants with stem cell transplant were reported in this outcome measure.
Time Frame: as for outcome 18
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 516 | 71
Participants | 125 | 26

30. Primary Outcome: Absolute Value of Hemoglobin Before Treatment Line
Description: Absolute value of hemoglobin before start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: Up to 48 hours before each treatment cycle till the end of treatment, disease progression and/or death from any cause; data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for the outcome measure. Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 470 | 59
Grams per deciliter
  LOT1 | 8.3 (1.7) | 9.2 (2.2)
  LOT2: number analyzed (Participants) | 236 | 42
  LOT2 | 9.2 (1.8) | 10.4 (2.2)
  LOT3: number analyzed (Participants) | 119 | 23
  LOT3 | 9.3 (2.1) | 9.9 (2.3)
  LOT4: number analyzed (Participants) | 43 | 10
  LOT4 | 9.2 (1.5) | 9.4 (2.2)
  LOT5-LOT7: number analyzed (Participants) | 26 | 6
  LOT5-LOT7 | 9.5 (2.2) | 9.9 (1.7)

31. Primary Outcome: Absolute Value of Hemoglobin After Start of Treatment Line
Description: Absolute value of hemoglobin after start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: After start of treatment until end of treatment, disease progression, death or loss of follow-up (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 416 | 55
Grams per deciliter
  LOT1 | 8.3 (1.6) | 10.0 (2.2)
  LOT2: number analyzed (Participants) | 232 | 42
  LOT2 | 8.7 (1.6) | 9.3 (2.3)
  LOT3: number analyzed (Participants) | 110 | 23
  LOT3 | 8.9 (2.1) | 9.5 (2.3)
  LOT4: number analyzed (Participants) | 50 | 10
  LOT4 | 8.6 (1.4) | 8.5 (1.7)
  LOT5-LOT7: number analyzed (Participants) | 20 | 5
  LOT5-LOT7 | 8.7 (1.6) | 9.2 (2.0)

32. Primary Outcome: Absolute Value of White Blood Cell Count Before Treatment Line
Description: Absolute value of white blood cell count before start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: as for outcome 30
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies total number of participants. 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: 10^9cells per Liter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 471 | 59
10^9cells per Liter
  LOT1 | 41.7 (168.6) | 35.7 (58.1)
  LOT2: number analyzed (Participants) | 236 | 42
  LOT2 | 12.6 (33.6) | 26.8 (48.4)
  LOT3: number analyzed (Participants) | 120 | 23
  LOT3 | 17.4 (34.0) | 26.4 (58.6)
  LOT4: number analyzed (Participants) | 43 | 10
  LOT4 | 7.9 (13.7) | 32.4 (69.3)
  LOT5-LOT7: number analyzed (Participants) | 26 | 6
  LOT5-LOT7 | 15.7 (39.3) | 17.0 (29.8)

33. Primary Outcome: Absolute Value of White Blood Cell Count After Start of Treatment Line
Description: Absolute value of white blood cell count after start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9cells per Liter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 416 | 55
10^9cells per Liter
  LOT1 | 7.8 (20.4) | 6.4 (6.7)
  LOT2: number analyzed (Participants) | 232 | 42
  LOT2 | 6.7 (18.3) | 10.7 (32.4)
  LOT3: number analyzed (Participants) | 110 | 22
  LOT3 | 16.3 (70.2) | 7.9 (18.2)
  LOT4: number analyzed (Participants) | 50 | 10
  LOT4 | 12.0 (40.7) | 4.9 (9.3)
  LOT5-LOT7: number analyzed (Participants) | 20 | 5
  LOT5-LOT7 | 6.8 (13.0) | 3.1 (2.3)

34. Primary Outcome: Absolute Neutrophil Count (ANC) Before Treatment Line
Description: Absolute value of neutrophil count before start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: Up to 1 week before treatment initiation; data collected and observed retrospectively over 11 months
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9cells per Liter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 432 | 57
10^9cells per Liter
  LOT1 | 5.0 (21.0) | 4.5 (6.5)
  LOT2: number analyzed (Participants) | 214 | 40
  LOT2 | 6.3 (13.7) | 5.7 (9.3)
  LOT3: number analyzed (Participants) | 110 | 21
  LOT3 | 8.8 (20.1) | 2.1 (2.0)
  LOT4: number analyzed (Participants) | 43 | 9
  LOT4 | 11.0 (23.8) | 1.9 (2.1)
  LOT5-LOT7: number analyzed (Participants) | 25 | 6
  LOT5-LOT7 | 15.1 (31.4) | 3.7 (2.3)

35. Primary Outcome: Absolute Neutrophil Count (ANC) After Start of Treatment Line
Description: Absolute value of neutrophil count after start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^9cells per Liter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 376 | 52
10^9cells per Liter
  LOT1 | 4.1 (10.5) | 6.8 (18.7)
  LOT2: number analyzed (Participants) | 208 | 40
  LOT2 | 4.9 (13.9) | 4.4 (9.7)
  LOT3: number analyzed (Participants) | 103 | 19
  LOT3 | 7.4 (19.4) | 1.9 (2.8)
  LOT4: number analyzed (Participants) | 45 | 8
  LOT4 | 12.4 (28.2) | 13.9 (27.5)
  LOT5-LOT7: number analyzed (Participants) | 19 | 5
  LOT5-LOT7 | 18.5 (32.4) | 2.1 (2.2)

36. Primary Outcome: Absolute Value of Blast Count Before Treatment Line
Description: Absolute value of blast count before start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: Up to 1 week before treatment initiation; data collected and observed retrospectively over 11 months
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percentage of blast cells
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 416 | 52
Percentage of blast cells
  LOT1 | 37.5 (33.4) | 36.4 (35.0)
  LOT2: number analyzed (Participants) | 207 | 31
  LOT2 | 12.0 (26.1) | 16.9 (30.0)
  LOT3: number analyzed (Participants) | 103 | 20
  LOT3 | 22.4 (35.8) | 20.4 (30.5)
  LOT4: number analyzed (Participants) | 34 | 7
  LOT4 | 11.2 (25.8) | 12.7 (27.7)
  LOT5-LOT7: number analyzed (Participants) | 17 | 6
  LOT5-LOT7 | 30.8 (35.2) | 14.7 (35.9)

37. Primary Outcome: Absolute Value of Blast Count After Start of Treatment Line
Description: Absolute value of blast count after start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percentage of blast cells
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 367 | 42
Percentage of blast cells
  LOT1 | 7.7 (19.8) | 7.2 (20.8)
  LOT2: number analyzed (Participants) | 205 | 34
  LOT2 | 6.9 (19.0) | 11.9 (28.5)
  LOT3: number analyzed (Participants) | 95 | 17
  LOT3 | 7.6 (21.9) | 13.6 (29.1)
  LOT4: number analyzed (Participants) | 38 | 9
  LOT4 | 9.2 (22.4) | 0.7 (2.0)
  LOT5-LOT7: number analyzed (Participants) | 11 | 5
  LOT5-LOT7 | 13.0 (23.0) | 0 (0)

38. Primary Outcome: Absolute Value of Platelets Count Before Treatment Line
Description: Absolute value of platelet count before start of treatment according to each line of treatment was reported in this outcome measure.
Time Frame: Up to 1 week before treatment initiation; data collected and observed retrospectively over 11 months
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 471 | 59
10^3 cells per microliter
  LOT1 | 68613 (75931) | 69220 (80225)
  LOT2: number analyzed (Participants) | 236 | 42
  LOT2 | 153362 (141776) | 115181 (110273)
  LOT3: number analyzed (Participants) | 119 | 23
  LOT3 | 112035 (120858) | 91565 (95696)
  LOT4: number analyzed (Participants) | 43 | 10
  LOT4 | 143263 (122895) | 69100 (96956)
  LOT5-LOT7: number analyzed (Participants) | 26 | 6
  LOT5-LOT7 | 101231 (113248) | 77200 (60318)

39. Primary Outcome: Absolute Value of Platelets Count After Start of Treatment Line
Description: Absolute value of platelet count after start of treatment according to different treatment lines were reported.
Time Frame: as for outcome 31
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 415 | 55
10^3 cells per microliter
  LOT1 | 105713 (153196) | 128894 (101555)
  LOT2: number analyzed (Participants) | 232 | 42
  LOT2 | 99613 (108309) | 78298 (79402)
  LOT3: number analyzed (Participants) | 109 | 23
  LOT3 | 75496 (77934) | 88996 (121220)
  LOT4: number analyzed (Participants) | 50 | 10
  LOT4 | 60340 (8533) | 39225 (12088)
  LOT5-LOT7: number analyzed (Participants) | 20 | 5
  LOT5-LOT7 | 93184 (320836) | 71300 (75856)

40. Secondary Outcome: Number of Participants With Molecular Test Performed
Description: Number of participants with different molecular test KGB, Fluorescence in situ hybridization (FISH), Reverse transcription polymerase chain reaction (RT-PCR), Next-generation sequencing (NGS), Array Comparative Genomic Hybridization (ACGH), Other performed were reported.
Time Frame: At diagnosis (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 427 | 65
Participants
  KGB | 381 | 52
  FISH | 112 | 31
  RT-PCR | 247 | 40
  NGS | 33 | 1
  ACGH | 0 | 0
  Other | 23 | 3

41. Secondary Outcome: Number of Participants According to AML Translocation Results: AML Arm Only
Description: Number of participants according to different AML translocation were reported in this outcome measure.
Time Frame: From diagnosis until loss of follow-up or death (up to maximum of 94.6 months ); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Only newly AML participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 319
Participants
  t(8;21) | 22
  inv(16) | 26
  der(11q23) | 1
  t(6;9) | 1
  t(1;22) | 0
  t(7;11) | 1
  inv(3) | 4
  t(16;21) | 0
  del(7q) | 7
  Monosomy 7(-7) | 9
  Complex cytogenetics/Complex karyotypes | 40
  Other | 208

42. Secondary Outcome: Number of Participants According to Molecular Profile in Newly AML Arm
Description: Number of participants according to molecular profile were reported in this outcome measure.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 286
Participants
  ASXL1 | 1
  BCOR | 2
  CEBPA | 13
  CSF3R | 1
  DNMT3A | 9
  EZH2 | 1
  IDH1 | 6
  IDH2 | 3
  KIT | 8
  KRAS | 1
  NPM1 | 66
  NRAS | 4
  PTPN11 | 1
  RUNX1 | 16
  SF3B1 | 0
  SRSF2 | 2
  STAG2 | 1
  TET2 | 4
  TP53 | 5
  U2AF1 | 0
  ZRSR2 | 0
  FLT3 | 94
  MLL-PTD | 3
  Other | 125

43. Secondary Outcome: Number of Participants According to AML WHO Classification: AML Arm Only
Description: Number of participants according to AML WHO classification were reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 391
Participants
  AML with recurrent genetic abnormalities | 28
  AML with t(8;21)(q22;q22.1);RUNX1 | 19
  AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22);CBFB | 28
  APL with PML | 0
  AML with t(9;11)(p21.3;q23.3);MLLT3 | 2
  AML with t(6;9)(p23;q34.1);DEK | 1
  AML with inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2); GATA2, MECOM | 3
  AML (megakaryoblastic) with t(1;22)(p13.3;q13.3);RBM15 | 0
  Provisional entity: AML with BCR | 0
  AML with mutated NPM1 | 36
  AML with biallelic mutations of CEBPA | 3
  Provisional entity: AML with mutated RUNX1 | 3
  AML with myelodysplasia | 27
  Therapy | 1
  AML, NOS | 240

44. Secondary Outcome: Number of Participants According to ALL WHO Classification: R/R B-cell ALL Arm Only
Description: Number of participants according to ALL WHO classification were reported in this outcome measure.
Time Frame: At diagnosis (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Only R/R B-cell ALL participants were to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 56
Participants
  B-lymphoblastic leukemia/lymphoma, NOS | 30
  B-lymphoblastic leukemia/lymphoma with recurrent genetic abnormalities | 0
  B-lymphoblastic leukemia/lymphoma with t(9;22)(q34.1;q11.2);BCR-ABL1 | 17
  B-lymphoblastic leukemia/lymphoma with t(v;11q23.3);KMT2A rearranged | 3
  B-lymphoblastic leukemia/lymphoma with t(12;21)(p13.2;q22.1); ETV6-RUNX1 | 0
  B-lymphoblastic leukemia/lymphoma with hyperdiploidy | 1
  B-lymphoblastic leukemia/lymphoma with hypodiploidy | 1
  B-lymphoblastic leukemia/lymphoma with t(5;14)(q31.1;q32.3) IL3-IGH | 0
  B-lymphoblastic leukemia/lymphoma with t(1;19)(q23;p13.3);TCF3-PBX1 | 0
  Provisional entity: B-lymphoblastic leukemia/lymphoma, BCR-ABL1-like | 4
  Provisional entity: B-lymphoblastic leukemia/lymphoma with iAMP21 | 0

45. Secondary Outcome: Number of Participants According to Immunophenotyping Results for AML Arm Only
Description: Number of participants according to immunophenotyping assessment results were reported for AML arm in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 468
Participants
  AML_IP_RES | 7
  cCD3 | 5
  cCD79a | 9
  MPO | 239
  CD34 | 316
  CD3 | 9
  CD4 | 43
  CD5 | 3
  CD7 | 119
  CD8 | 6
  TdT | 2
  CD10 | 14
  CD19 | 30
  CD20 | 6
  CD13 | 364
  CD33 | 354
  CD14 | 49
  CD36 | 87
  HLADR | 376
  glycophorin A | 1
  CD41 | 1
  CD61 | 4
  CD117 | 400
  Other | 327

46. Secondary Outcome: Number of Participants According to Immunophenotyping Results for R/R B-cell ALL
Description: Number of participants according to immunophenotyping assessment results were reported for R/R B-cell ALL arm in this outcome measure.
Time Frame: At diagnosis (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 20
Participants
  CD19 | 18
  CD20 | 6
  CD22 | 11
  CD79a | 9
  HLA Dr | 6
  TdT | 7
  CD10 | 17
  CD34 | 18
  CD45 | 11
  Cytoplasmic IgM | 1
  Other | 9

47. Secondary Outcome: Number of Participants According to Molecular Profile in R/R B-cell ALL
Description: Number of participants according to molecular profile in R/R B-cell ALL were reported.
Time Frame: At diagnosis (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 53
Participants
  B-cell immunoglobulin gene rearrangement | 1
  inv(16) | 0
  der(11q23) | 21
  t(6;9) | 0
  t(4;11) | 3
  Other | 28

48. Secondary Outcome: Number of Participants According to ALL Cytogenetic Risk Classification: R/R B-cell ALL Arm Only
Description: A good prognosis means that there was a high chance of recovery or healing. Intermediate prognosis was a term used to describe the likelihood of recovery or survival from a disease or condition that was neither favorable nor unfavorable. A poor prognosis refers to an estimation that there was a low chance of recovery from a disease.
Time Frame: At diagnosis (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 52
Participants
  Good prognosis | 1
  Intermediate prognosis | 16
  Poor prognosis | 29
  Undetermined prognosis | 6

49. Secondary Outcome: Number of Participants According to AML Cytogenetic Risk Classification Based on 2017 European Leukemia Net (ELN)
Description: Number of participants according to AML Cytogenetic Risk Classification Based on 2017 European Leukemia Net (ELN)" under favorable (indicates a low probability or impact of adverse outcomes), intermediate (associated with moderate changes) and Poor/ Adverse (occurrence of a risk was high and the impact of the risk is severe) were reported.
Time Frame: as for outcome 13
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML
Number analyzed (Participants) | 373
Participants
  Favorable | 85
  Intermediate | 179
  Poor/Adverse | 109

50. Secondary Outcome: Number of Participants According to Drug Regimen Prescribed Since Diagnosis of de Novo ALL in R/R B-cell ALL
Description: A regimen could be a treatment that consisted of one or combined (two or more) drugs. Number of participants according to drug regimen prescribed for R/R B-cell ALL is reported. Hyper- CVAD (hyper fractionated cyclophosphamide, vincristine, doxorubicin, and prednisolone), German multicenter ALL (GMALL), GRAAL, Berlin-Frankfurt-Münster (BFM), Inotuzumab, Blinatumomab Chimeric antigen receptor T-cell therapies (CAR-T), Tyrosine kinase inhibitors (TKI), FLAG (fludarabine + high-dose cytarabine + G-CSF), FLAG-IDA Regimen (Fludarabine, Cytarabine, Idarubicin and G-CSF). The initial diagnosis of acute leukemia could have been before 01-Jan-2015.
Time Frame: From the diagnosis for de novo ALL diagnosis date to study enrolment date (anytime between 2001-2014 approximately 13 years); data collected and observed retrospectively over 11 months
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | R/R B-cell ALL
Number analyzed (Participants) | 65
Participants
  Hyper-CVAD (since de novo ALL diagnose date) | 13
  GMALL (since de novo ALL diagnose date) | 0
  GRAAL (since de novo ALL diagnose date) | 7
  BFM (since de novo ALL diagnose date) | 16
  Inotuzumab (since de novo ALL diagnose date) | 0
  Blinatumomab (since de novo ALL diagnose date) | 1
  Car T-cell (since de novo ALL diagnose date) | 0
  TKI inhibitor (since de novo ALL diagnose date) | 5
  FLAG (since de novo ALL diagnose date) | 0
  FLAG-IDA (since de novo ALL diagnose date) | 2
  Other (since de novo ALL diagnose date) | 28

51. Secondary Outcome: Time From Start of First-Line Treatment to Start of the Adverse Event
Description: Time from start of first line treatment to start of the adverse event were reported. An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From start of 1st line treatment until Adverse Event (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 3 | 1
Months | 56.0 (15.8) | 39.5 (28.0)

52. Secondary Outcome: Number of Clinical Events
Description: Number of clinical events were reported in this outcome measure.
Time Frame: From diagnosis until end of treatment, disease progression, death or loss of follow-up (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, 'Number Analyzed' signifies events evaluable for the specified rows.
Measure: Number; unit: Events
Units Other Than Participants: clinical events
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Number analyzed (clinical events) | 1220 | 218
Events
  Hematological toxicities | 317 | 86
  Hepatotoxicity | 5 | 7
  Gastrointestinal toxicities | 86 | 17

53. Secondary Outcome: Event Free Survival (EFS)
Description: EFS =time since treatment initiation until failure to achieve complete remission (CR) or disease progression (PD) after CR, or death from any cause. Participants not known to have any of these events were censored on the date they were last examined, study enrollment, last contact, whichever came later.CR=participants response to treatment according to the medical chart. AML CR =no physical signs of leukemia, bone marrow with active hematopoiesis, <5% bone marrow blasts and more than 1* 10^9 cells/l granulocytes and more than 100* 10^9 cells/l platelets in the blood and no circulating leukemic blasts or evidence of extramedullary leukemia), PD=according to medical chart and accompanied by a decline in absolute neutrophil count (ANC) and platelets and increased transfusion requirement and decline in performance status or increase in symptoms.
Time Frame: From start of treatment until failure to achieve CR, PD or death or censoring date (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 508 | 79
Months | 1.5 [1.4 to 1.7] | 1.8 [1.4 to 2.7]

54. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of diagnosis or treatment until date of death due to any cause. If there was no death, the participants were censored at last visit or contact, whichever came later.
Time Frame: From start of treatment until disease progression, loss of follow-up or death (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 517 | 71
Months | 10.6 [8.6 to 12.2] | 19.2 [15.4 to 32.0]

55. Secondary Outcome: Secondary: Percentage of Participants Alive at 1,3 and 5 Years Since Treatment Initiation
Description: Percentage of participants alive at 1,3 and 5 years since treatment initiation were reported in this outcome measure.
Time Frame: 1, 3 and 5 years since treatment initiation; data collected and observed retrospectively over 11 months
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 517 | 71
Percentage of participants
  1 year | 47.7 | 67.6
  3 years | 28.0 | 35.2
  5 years | 24.5 | 19.7

56. Secondary Outcome: Relapse Free Survival-Newly Diagnosed AML Participants Only
Description: Relapse was a deterioration in health status after an improvement. Relapse free survival was considered as date of achievement of a remission until the date of relapse or death from any cause; participants not known to have relapsed or died at last follow-up were censored on the date they were last examined. CR=a participant's response to treatment according to the medical chart. Usually, AML complete remission defined as no physical signs of leukemia, bone marrow with active hematopoiesis, <5% bone marrow blasts and more than 1* 10^9 cells/L granulocytes and more than 100* 10^9 cells/L platelets in the blood and no circulating leukemic blasts or evidence of extramedullary leukemia.
Time Frame: From date of remission until relapse or death or censoring date (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: as for outcome 41
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly AML
Number analyzed (Participants) | 383
Months | 3.9 [3.0 to 5.0]

57. Secondary Outcome: Number of Participants According to Treatment Response
Description: Complete remission-response (CR) defined as no physical signs of leukemia, bone marrow with active hematopoiesis, <5% bone marrow blasts and more than 1×109/l granulocytes and more than 100×109/l platelets in blood and no circulating leukemic blasts or evidence of extramedullary leukemia. Complete response with incomplete blood count recovery (CRi): also known as CR with incomplete hematologic recovery, participant's response to treatment according to medical chart. Partial remission: participant's response to treatment according to medical chart. All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; decrease of pretreatment bone marrow blast percentage by at least 50%. Disease progression: >25% increase in sum of longest diameter of target lesions compared to baseline. Refractory disease: according to medical chart. No CR after 2 courses of intensive induction treatment; excluding participants with death in aplasia or death due to indeterminate cause.
Time Frame: as for outcome 54
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 456 | 68
Participants
  Complete remission-response (LOT1) | 190 | 24
  Complete remission-response with incomplete hematological-count recovery (LOT1) | 16 | 7
  Partial remission-response (LOT1) | 27 | 5
  Progressive disease (LOT1) | 33 | 9
  Refractory disease (LOT1) | 142 | 19
  Relapsed from CR or CRi or recurrent disease (LOT1) | 12 | 3
  Other (LOT1) | 36 | 1
  Complete remission-response (LOT2): number analyzed (Participants) | 259 | 49
  Complete remission-response (LOT2) | 129 | 12
  Complete remission-response with incomplete hematological-count recovery (LOT2): number analyzed (Participants) | 259 | 49
  Complete remission-response with incomplete hematological-count recovery (LOT2) | 11 | 5
  Partial remission-response (LOT2): number analyzed (Participants) | 259 | 49
  Partial remission-response (LOT2) | 12 | 4
  Progressive disease (LOT2): number analyzed (Participants) | 259 | 49
  Progressive disease (LOT2) | 19 | 5
  Refractory disease (LOT2): number analyzed (Participants) | 259 | 49
  Refractory disease (LOT2) | 58 | 18
  Relapsed from CR or CRi or recurrent disease (LOT2): number analyzed (Participants) | 259 | 49
  Relapsed from CR or CRi or recurrent disease (LOT2) | 14 | 2
  Other (LOT2): number analyzed (Participants) | 259 | 49
  Other (LOT2) | 16 | 3
  Complete remission-response (LOT3): number analyzed (Participants) | 133 | 25
  Complete remission-response (LOT3) | 54 | 3
  Complete remission-response with incomplete hematological-count recovery (LOT3): number analyzed (Participants) | 133 | 25
  Complete remission-response with incomplete hematological-count recovery (LOT3) | 2 | 1
  Partial remission-response (LOT3): number analyzed (Participants) | 133 | 25
  Partial remission-response (LOT3) | 2 | 0
  Progressive disease (LOT3): number analyzed (Participants) | 133 | 25
  Progressive disease (LOT3) | 9 | 4
  Refractory disease (LOT3): number analyzed (Participants) | 133 | 25
  Refractory disease (LOT3) | 47 | 12
  Relapsed from CR or CRi or recurrent disease (LOT3): number analyzed (Participants) | 133 | 25
  Relapsed from CR or CRi or recurrent disease (LOT3) | 8 | 0
  Other (LOT3): number analyzed (Participants) | 133 | 25
  Other (LOT3) | 11 | 5
  Complete remission-response (LOT4): number analyzed (Participants) | 56 | 11
  Complete remission-response (LOT4) | 27 | 3
  Complete remission-response with incomplete hematological-count recovery (LOT4): number analyzed (Participants) | 56 | 11
  Complete remission-response with incomplete hematological-count recovery (LOT4) | 0 | 0
  Partial remission-response (LOT4): number analyzed (Participants) | 56 | 11
  Partial remission-response (LOT4) | 2 | 0
  Progressive disease (LOT4): number analyzed (Participants) | 56 | 11
  Progressive disease (LOT4) | 6 | 0
  Refractory disease (LOT4): number analyzed (Participants) | 56 | 11
  Refractory disease (LOT4) | 18 | 5
  Relapsed from CR or CRi or recurrent disease (LOT4): number analyzed (Participants) | 56 | 11
  Relapsed from CR or CRi or recurrent disease (LOT4) | 2 | 0
  Other (LOT4): number analyzed (Participants) | 56 | 11
  Other (LOT4) | 1 | 3
  Complete remission-response (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Complete remission-response (LOT5-LOT7) | 8 | 4
  Complete remission-response with incomplete hematological-count recovery (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Complete remission-response with incomplete hematological-count recovery (LOT5-LOT7) | 2 | 0
  Partial remission-response (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Partial remission-response (LOT5-LOT7) | 0 | 0
  Progressive disease (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Progressive disease (LOT5-LOT7) | 3 | 0
  Refractory disease (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Refractory disease (LOT5-LOT7) | 8 | 2
  Relapsed from CR or CRi or recurrent disease (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Relapsed from CR or CRi or recurrent disease (LOT5-LOT7) | 1 | 0
  Other (LOT5-LOT7): number analyzed (Participants) | 25 | 6
  Other (LOT5-LOT7) | 3 | 0

58. Secondary Outcome: Number of Hospitalizations
Description: Number of hospitalizations were reported in this outcome measure. One participant could have more than one hospitalization.
Time Frame: From diagnosis until end of treatment, loss of follow-up or death (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Hospitalizations
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Hospitalizations | 880 | 128

59. Secondary Outcome: Reason for Hospitalization
Description: Reason for hospitalizations according to reasons such as ALL-AML treatment, adverse events were reported. One participant could have more than one reason for hospitalization.
Time Frame: as for outcome 58
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Hospitalization
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Hospitalization
  ALL-AML Treatment | 1064 | 236
  Adverse events | 20 | 4
  Other | 559 | 134

60. Secondary Outcome: Duration in Intensive Care Unit
Description: Mean duration in intensive care unit were reported in this outcome measure.
Time Frame: as for outcome 58
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 280 | 46
Days | 9.1 (11.4) | 11.4 (12.7)

61. Secondary Outcome: Number of Procedures
Description: Different clinical procedures were reported. One participant could have more than one procedure.
Time Frame: as for outcome 58
Population: as for outcome 31
Measure: Number; unit: Procedures
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Procedures
  Surgery | 60 | 8
  Image exams | 1187 | 172
  Laboratory exams | 1494 | 311
  Blood transfusions | 1128 | 162
  Associated treatments for infections | 1062 | 153
  Use of mechanical ventilation | 141 | 18
  Use of parenteral feeding | 231 | 11
  Other | 70 | 19

62. Secondary Outcome: Number of Participants According to Surgery
Description: Number of participants according to type of surgery were reported in this outcome measure.
Time Frame: as for outcome 58
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 60 | 8
Participants
  Abcess | 9 | 0
  Catheter | 2 | 2
  Tracheostomy | 4 | 0
  Other | 45 | 6

63. Secondary Outcome: Number of Blood Transfusions
Description: Number and type of blood transfusions were reported in this outcome measure. One participant could have more than one blood transfusions.
Time Frame: as for outcome 58
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Blood transfusions
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Blood transfusions
  Platelet | 1032 | 121
  Plasma | 107 | 16
  Red blood cells | 1051 | 139
  Whole blood | 63 | 4
  Other | 3 | 1

64. Secondary Outcome: Number of Concomitant Medications
Description: Concomitant medication: drug treatment for comorbidities, supportive and prophylaxis therapies, or to treat adverse events.
Time Frame: as for outcome 58
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Medications
Units Other Than Participants: concomitant medication
Arm/Group | Newly AML | R/R B-cell ALL
Number analyzed (Participants) | 518 | 71
Number analyzed (concomitant medication) | 3343 | 501
Medications
  Vancomycin | 268 | 36
  Meropenem | 252 | 34
  Piperacillin; Tazobactam | 219 | 36
  Other | 2604 | 395

ADVERSE EVENTS:
Time Frame: From start of treatment until end of treatment, death or loss of follow-up (up to maximum of 94.6 months); data collected and observed retrospectively over 11 months
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Newly AML | R/R B-cell ALL
All-Cause Mortality (participants affected / at risk) | 392/518 | 60/71
Serious Adverse Events (participants affected / at risk) | 2/518 | 0/71
Other Adverse Events (participants affected / at risk) | 2/518 | 1/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newly AML (N=518) | R/R B-cell ALL (N=71)
Sepsis (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newly AML (N=518) | R/R B-cell ALL (N=71)
Renal Failure (Renal and urinary disorders) | 0 | 1
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT05166135/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT05166135/SAP_001.pdf